CLINICAL TRIAL: NCT00727298
Title: Post Marketing Surveillance Study of the Labeled Use of Remicade® (Infliximab) in Patients With Chronic Inflammatory Diseases
Brief Title: Post Marketing Surveillance Study of Remicade in Patients With Chronic Inflammatory Diseases (P04840)
Acronym: REMission
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P04840
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Psoriasis; Crohn's Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Psoriasis; Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab: Infliximab administered at a dose of 3-10 mg/kg at Week 0, Week 2, and Week 6, and every 4-8 weeks thereafter for 24 months for the treatment of chronic inflammatory disease.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab administered at a dose of 3-10 mg/kg at Week 0, Week 2, and Week 6, and every 4-8 weeks thereafter for 24 months for the treatment of chronic inflammatory disease.
  Other Names: Remicade; SCH 215596

SUMMARY:
This study will be performed to evaluate and document the safety and efficacy of infliximab (Remicade®) in the treatment of chronic inflammatory diseases in big cohorts in the daily routine practice of rheumatologists, gastroenterologists, and dermatologists.

DETAILED DESCRIPTION:
The study population was chosen from a non-probability sample.

The safety population consisted of all participants with at least one documented infusion of infliximab.

The evaluable population consisted of all participants that were >=18 years of age with a recorded indication for infliximab use, that had available baseline data, and with at least 3 infusions of infliximab within the first 16 weeks of the study. Baseline characteristics are provided for this population.

ELIGIBILITY:
Inclusion Criteria:

* Participants treated with infliximab by rheumatologists, gastroenterologists, and dermatologists for chronic inflammatory diseases, such as rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, psoriasis, or Crohn's disease.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants treated with infliximab by rheumatologists, gastroenterologists, and dermatologists for chronic inflammatory diseases, such as rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, psoriasis, or Crohn's disease.
Sampling Method: Non-Probability Sample
Enrollment: 4485 (Actual)
Dates: Start 2006-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 4485 total enrolled participants, 4465 received at least one infusion of infliximab and are included in the safety evaluation. 3228 of these participants were evaluable for all other study analyses.
Groups:
- Infliximab: Infliximab administered at a dose of 3-10 mg/kg administered at Week 0, Week 2, and Week 6, and every 4-8 weeks thereafter for 24 months for the treatment of chronic inflammatory disease.
Period: Overall Study
Arm/Group | Infliximab
Started | 4485
Completed | 3228
Not Completed | 1257

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 3228
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.9)
Sex/Gender, Customized [Number; unit: participants]
  Female | 1591
  Male | 1554
  Not Specified | 83

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing at Least One Adverse Event
Description: An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the treatment, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the treatment, was also an adverse event.
Time Frame: Baseline to Month 24
Population: The safety evaluable population consisted of all participants with that received at least one infusion of infliximab.
Measure: Number; unit: Participants
Groups:
- Infliximab 3-10 mg/kg: Infliximab administered at a dose of 3-10 mg/kg at Week 0, Week 2, and Week 6, and every 4-8 weeks thereafter for 24 months for the treatment of chronic inflammatory disease.
Arm/Group | Infliximab 3-10 mg/kg
Number analyzed (Participants) | 4465
Participants | 609

2. Secondary Outcome: Clinicians' Impression of Disease Severity From Baseline to Week 102
Description: Participant severity of disease was assessed at baseline, Week 6, Week 14, Week 22, Week 54, and Week 102 on the basis of the treating clinician's opinion of the participant being normal, not at all ill, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, or extreme severe illness. Each time point was compared to the previous visit.
Time Frame: Baseline, Week 6, Week 14, Week 22, Week 54, Week 102
Population: The efficacy evaluable population consisted of all participants with baseline data available that received at least 3 infusions of study drug within 14+2 weeks.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infliximab 3-10 mg/kg
Number analyzed (Participants) | 3228
Percentage of Participants
  Baseline - Not at all ill | 0.7
  Baseline - Borderline ill | 1.3
  Baseline - Mildly ill | 4.9
  Baseline - Moderately ill | 17.6
  Baseline - Markedly ill | 51.2
  Baseline - Severely ill | 21.0
  Baseline - Extreme severe illness | 2.8
  Week 6 - Not at all ill | 5.1
  Week 6 - Borderline ill | 10.5
  Week 6 - Mildly ill | 23.6
  Week 6 - Moderately ill | 27.7
  Week 6 - Markedly ill | 24.3
  Week 6 - Severely ill | 7.5
  Week 6 - Extreme severe illness | 1.1
  Week 14 - Not at all ill | 8.3
  Week 14 - Borderline ill | 14.2
  Week 14 - Mildly ill | 23.3
  Week 14 - Moderately ill | 26.1
  Week 14 - Markedly ill | 21.2
  Week 14 - Severely ill | 5.9
  Week 14 - Extreme severe illness | 0.8
  Week 22 - Not at all ill | 10.6
  Week 22 - Borderline ill | 14.8
  Week 22 - Mildly ill | 22.7
  Week 22 - Moderately ill | 25.5
  Week 22 - Markedly ill | 19.5
  Week 22 - Severely ill | 5.9
  Week 22 - Extreme severe illness | 0.8
  Week 54 - Not at all ill | 12.9
  Week 54 - Borderline ill | 16.3
  Week 54 - Mildly ill | 22.2
  Week 54 - Moderately ill | 23.3
  Week 54 - Markedly ill | 19.3
  Week 54 - Severely ill | 4.8
  Week 54 - Extreme severe illness | 1.0
  Week 102 - Not at all ill | 17.2
  Week 102 - Borderline ill | 16.5
  Week 102 - Mildly ill | 21.1
  Week 102 - Moderately ill | 22.2
  Week 102 - Markedly ill | 17.1
  Week 102 - Severely ill | 4.1
  Week 102 - Extreme severe illness | 1.3

3. Secondary Outcome: Clinicians' Impression of Therapeutic Efficacy
Description: Therapeutic efficacy was rated by the treating physician at each time point as moderate-to-clear improvement, no change, not assessable, mild-to-slight improvement, very good-to-full improvement, or worsened. Each time point was compared to the previous visit.
Time Frame: Week 6, Week 14, Week 22, Week 54, Week 102
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Infliximab 3-10 mg/kg
Number analyzed (Participants) | 3228
Percentage of Participants
  Week 6: Moderate-to-Clear Improvement | 34.8
  Week 6: Unchanged | 8.9
  Week 6: Not Assessable | 1.4
  Week 6: Mild-to-Slight Improvement | 17.4
  Week 6: Very Good-to-Full Improvement | 37.3
  Week 6: Worsened | 0.2
  Week 14: Moderate-to-Clear Improvement | 30.1
  Week 14: Unchanged | 9.9
  Week 14: Not Assessable | 1.5
  Week 14: Mild-to-Slight Improvement | 15.1
  Week 14: Very Good-to Full Improvement | 43.1
  Week 14: Worsened | 0.3
  Week 22: Moderate-to-Clear Improvement | 29.5
  Week 22: Unchanged | 11.3
  Week 22: Not Assessable | 1.9
  Week 22: Mild-to-Slight Improvement | 13.0
  Week 22: Very Good-to-Full Improvement | 43.9
  Week 22: Worsened | 0.3
  Week 54: Moderate-to-Clear Improvement | 27.0
  Week 54: Unchanged | 15.1
  Week 54: Not Assessable | 1.6
  Week 54: Mild-to-Slight Improvement | 9.3
  Week 54: Very Good-to-Full Improvement | 46.4
  Week 54: Worsened | 0.5
  Week 102: Moderate-to-Clear Improvement | 25.7
  Week 102: Unchanged | 16.3
  Week 102: Not Assessable | 1.7
  Week 102: Mild-to-Slight Improvement | 5.6
  Week 102: Very Good-to-Full Improvement | 50.0
  Week 102: Worsened | 0.6

ADVERSE EVENTS:
Description: The safety evaluable population consisted of all participants with that received at least one infusion of infliximab.
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 296/4465
Other Adverse Events (participants affected / at risk) | 0/4465
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=4465)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cadiovascular disorder (Cardiac disorders) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 10 (10)
Blindness transient (Eye disorders) | 1 (1)
Eyelid Oedema (Eye disorders) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Parathesia oral (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 6 (9)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 5 (5)
Condition aggravated (General disorders) | 2 (2)
Impaired healing (General disorders) | 2 (2)
Infusion related reaction (General disorders) | 28 (28)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sense of oppression (General disorders) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Anaphylactic reactions (Immune system disorders) | 3 (3)
Anaphylactic shock (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 16 (18)
Sarcoidosis (Immune system disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 2 (2)
Hepatitis B (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Purulence (Infections and infestations) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured ischium (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Antinuclear antibody increased (Investigations) | 2 (2)
Antinuclear antibody positive (Investigations) | 2 (2)
Blood pressure (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 9 (9)
Blood pressure decreased (Investigations) | 5 (5)
Blood pressure increased (Investigations) | 2 (2)
Blood pressure orthostatic (Investigations) | 2 (2)
DNA antibody positive (Investigations) | 1 (1)
Systemic lupus erythematosus disease activity index abnormal (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nodular fasciitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Neuritis (Nervous system disorders) | 1 (1)
Parathesia (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 5 (5)
Completed suicide (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (36)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritis generalised (Skin and subcutaneous tissue disorders) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Uticaria (Skin and subcutaneous tissue disorders) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Abscess drainage (Surgical and medical procedures) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 1 (1)
Bunion operation (Surgical and medical procedures) | 1 (1)
Bursa removal (Surgical and medical procedures) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Elbow operation (Surgical and medical procedures) | 1 (1)
Foot operation (Surgical and medical procedures) | 3 (3)
Glaucoma surgery (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 3 (3)
Hip surgery (Surgical and medical procedures) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 3 (3)
Intraocular lens implant (Surgical and medical procedures) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 2 (2)
Limb operation (Surgical and medical procedures) | 1 (1)
Polypectomy (Surgical and medical procedures) | 1 (1)
Proctocolectomy (Surgical and medical procedures) | 1 (1)
Rheumatoid nodule removal (Surgical and medical procedures) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 1 (1)
Sigmoidectomy (Surgical and medical procedures) | 3 (3)
Surgery (Surgical and medical procedures) | 3 (3)
Synovectomy (Surgical and medical procedures) | 1 (1)
Thyroid operation (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 10 (10)
Hypertension (Vascular disorders) | 6 (6)
Hypertensive crisis (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No